CLINICAL TRIAL: NCT03284177
Title: A Multicenter, Open-label Trial to Investigate the Safety of C13-CAC and the Relationship Among C13-CAC Breath Test, Gastric pH, and the Improvement of Symptoms in PPI Resistant GERD Patients
Brief Title: A Trial of C13-CAC Breath Test in PPI Resistant GERD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 334-103-00001; JapicCTI-173713 (Registry Identifier: Japic Clinical Trials Information)
Record Dates: First submitted 2017-09-11; First posted 2017-09-15 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Calcium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C13-CAC (Experimental)
  Interventions: Drug: Calcium (13C)Carbonate; Drug: Gastric acid inhibitors; Other: Gastric pH monitoring

INTERVENTIONS:
Drug: Calcium (13C)Carbonate — C13-CAC breath test containing Calcium (13C) Carbonate was performed twice under fasting conditions.
Drug: Gastric acid inhibitors — Gastric acid inhibitor was orally administrated once daily for 4weeks after first C13-CAC breath test.
Other: Gastric pH monitoring — Gastric pH monitoring was performed once under fasting condition.

SUMMARY:
To investigate the safety of C13-CAC and the relationship among C13-CAC breath test, gastric pH, and the improvement of symptoms by switching PPI in PPI resistant GERD patients

ELIGIBILITY:
Inclusion Criteria:

* GERD patients who have been judged to require additional treatment to improve their symptoms by investigator or subinvestigator.

Exclusion Criteria:

* Patients suspected to have hypothyroidism or hyperparathyroidism.
* Patients with hypercalcemia
* Patients with a history of gastric or duodenal surgery.
* Patients who have received the eradication therapy of Helicobacter pylori within six months prior to participation of the study.
* Patients with a prior or current history of Zollinger-Ellison syndrome.
* Patients with a history of surgery or treatment affecting gastroesophageal reflux.
* Patients who have been diagnosed with acute upper gastrointestinal bleeding or active gastric or duodenal ulcer within 30 days prior to participation of the study.
* Patients with serious central nervous system disorders, cardiovascular disease, pulmonary disease, hepatic disease, renal disease, metabolic disease, gastrointestinal disorders, urinary disorders, endocrine disease, or blood dyspraxia.
* Patients scheduled for surgery requiring hospitalization or required surgery during the study period.
* Patients who have had either a prior or current history of chest pain due to heart disease or with chest pain suspected to have caused by heart disease within one year prior to participation of the study.

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
13CO2 concentration in expired air. | 5，10，15，20，25 and 30 minutes after C13-CAC administration.
  Sensitivity and specificity of 13CO2 concentration in expired air for improvement of symptoms.

SECONDARY OUTCOMES:
Gastric pH | 1 hour prior to C13-CAC administration
  Sensitivity and specificity of mean gastric pH for improvement of symptoms.

CONTACTS AND LOCATIONS:
Locations (13):
- Japan (13):
  - Akita University Hospital, Akita
  - National Hospital Organization Hakodate Hospital, Hakodate
  - Shimane University Hospital, Izumo
  - Kawasaki Medical School General Medical Center, Kurashiki
  - Kawasaki Medical School Hospital, Kurashiki
  - National Hospital Organization Matsumoto Medical Center, Matsumoto
  - Hyogo College Of Medicine College Hospital, Nishinomiya
  - Osaka Saiseikai Nakatsu Hospital, Osaka
  - Center Hospital of the National Center for Global Health and Medicine, National Research and Development Agency, Tokyo
  - Hiratsuka stomach and intestines Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - National Hospital Organization Yokohama Medical Center, Yokohama
  - Yokohama City University Hospital, Yokohama

IPD SHARING:
Plan to Share IPD: No